CLINICAL TRIAL: NCT05432271
Title: A Large-scale, Long-term, Randomized Trial of Nutrition Labeling Interventions
Brief Title: Online Food and Beverage Labels and Vending Machine Selections
Acronym: VLO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 850263; R01DK113307 (NIH)
Record Dates: First submitted 2022-06-15; First posted 2022-06-27 (Actual); Results first posted 2023-12-20 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Food Preferences; Obesity; Weight Gain
Keywords: food labeling; sugar-sweetened beverages; eating; drinking; choice behavior
MeSH Terms: conditions — Food Preferences; Obesity; Weight Gain

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to 1 of 5 front-of-package labeling arms with equal probability: Participants will complete two vending machine choice tasks with their assigned labels shown (one for beverages, one for snack foods, in random order). For each choice task, participants will be asked to select 1 item they most wish to purchase. We will incentivize truthful responding by instructing participants that they could be randomly selected to have their choice delivered to them. We will record participants' selections and match these to nutrition information.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Control (Active Comparator): Calorie labels shown on front of product packaging
  Interventions: Behavioral: Exposure to calorie information
- Green labels (Experimental): Green label added to front of product packaging for healthy products; no additional labels shown for "less healthy" products
  Interventions: Behavioral: Exposure to calorie information; Behavioral: Exposure to healthy labels only
- Traffic light labels (Experimental): Red/yellow/green labels added to front of product packaging for less healthy/moderately healthy/healthy products, respectively
  Interventions: Behavioral: Exposure to calorie information; Behavioral: Exposure to healthiness information
- Physical activity calorie equivalent labels (Experimental): Labels added to front of product packaging that display products' calorie content in terms of physical activity required to burn those calories
  Interventions: Behavioral: Exposure to calorie information; Behavioral: Exposure to physical activity equivalents
- "High in" nutrient warning labels (Experimental): Labels added to front of product packaging that signal when the product exceeds thresholds for sugar, sodium, saturated fat, or calorie content
  Interventions: Behavioral: Exposure to calorie information; Behavioral: Exposure to "high in" nutrient warning labels

INTERVENTIONS:
Behavioral: Exposure to calorie information — Calories for all beverages and foods
Behavioral: Exposure to healthy labels only — Green labels only for beverages and foods scored as healthy
  Arms: Green labels
Behavioral: Exposure to healthiness information — All beverages and foods labeled as either healthy (green), moderately healthy (yellow), or less healthy (red)
  Arms: Traffic light labels
Behavioral: Exposure to physical activity equivalents — All beverages and foods labeled with physical activity required to burn their calories
  Arms: Physical activity calorie equivalent labels
Behavioral: Exposure to "high in" nutrient warning labels — Warning labels only for beverages and foods that exceed the thresholds for sugar, sodium, saturated fat, or calorie content
  Arms: "High in" nutrient warning labels

SUMMARY:
The aim of this study is to compare the impact of 5 different types of front of package (FOP) food and beverage labels: 1) calorie labels [control], 2) green labels on healthy foods, 3) red/yellow/green labels on less healthy/moderately healthy/healthy foods, 4) physical activity calorie equivalent labels, and 5) "High in" nutrient warning labels) on consumers' beverage and snack selections.

DETAILED DESCRIPTION:
This project involves an online randomized experiment. We are working with an external survey company that will recruit 8,000 participants to complete an online survey in which they will be randomized to one of the five different label conditions: 1) calorie labels (control condition); 2) single green traffic light labels (on healthy foods); 3) multiple traffic light labels (red traffic light labels applied to less healthy foods, yellow applied to moderately healthy foods, and green on healthy foods); 4) physical activity labels (calorie content displayed in terms of physical activity equivalents); 5) "High in" warnings (applied to all products exceeding thresholds for calories, saturated fat, sugar, or sodium content). Participants will be instructed to select products to purchase in a mock vending machine. After purchasing their products, they will be asked to answer questions about their perceptions of the different labels.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be US adults
* Ages 18 or older
* With an over-sample of adults with lower educational attainment (some college or less)

Exclusion Criteria:

* Younger than 18
* Non-US
* Educational quota filled

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8145 (Actual)
Dates: Start 2022-11-16 (Actual); Primary Completion 2022-12-03 (Actual); Study Completion 2022-12-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christina A Roberto, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
In the consenting process, participants agreed that de-identified data produced from this project may be distributed for future research studies without additional informed consent. After analysis, we will upload the de-identified data to ResearchBox for public sharing.
Supporting Information: SAP
Time Frame: Starting 6 months after publication
Access Criteria: Public

REFERENCES:
- [Derived] Grummon AH, Gibson LA, Musicus AA, Stephens-Shields AJ, Hua SV, Roberto CA. Effects of 4 Interpretive Front-of-Package Labeling Systems on Hypothetical Beverage and Snack Selections: A Randomized Clinical Trial. JAMA Netw Open. 2023 Sep 5;6(9):e2333515. doi: 10.1001/jamanetworkopen.2023.33515. PMID 37703015

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control | Green Labels | Traffic Light Labels | Physical Activity Calorie Equivalent Labels | "High in" Nutrient Warning Labels
Started | 1627 | 1639 | 1623 | 1633 | 1623
Completed | 1627 | 1639 | 1623 | 1633 | 1623
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Participants were excluded from analysis if a) they requested their data be excluded after being debriefed about the purpose of the study or b) they finished the survey too quickly (i.e., faster than 191.2 seconds which was 1/3 of the median completion time in a soft launch of the survey).
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Green Labels | Traffic Light Labels | Physical Activity Calorie Equivalent Labels | "High in" Nutrient Warning Labels | Total
Number analyzed (Participants) | 1593 | 1587 | 1588 | 1590 | 1587 | 7945
Age, Customized [Count of Participants; unit: Participants]
  Age in years: 18-29 | 310 | 311 | 324 | 317 | 343 | 1605
  Age in years: 30-44 | 419 | 382 | 402 | 408 | 408 | 2019
  Age in years: 45-59 | 426 | 394 | 385 | 374 | 389 | 1968
  Age in years: >=60 | 438 | 500 | 477 | 491 | 447 | 2353
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender: Female | 814 | 799 | 825 | 844 | 796 | 4078
  Gender: Male | 757 | 773 | 746 | 729 | 774 | 3779
  Gender: Nonbinary or another gender | 22 | 15 | 17 | 17 | 17 | 88
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 295 | 235 | 270 | 246 | 251 | 1297
  Not Hispanic or Latino | 1298 | 1352 | 1318 | 1344 | 1335 | 6647
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 26 | 27 | 25 | 24 | 17 | 119
  Asian | 30 | 32 | 42 | 50 | 42 | 196
  Native Hawaiian or Other Pacific Islander | 9 | 6 | 7 | 5 | 9 | 36
  Black or African American | 193 | 206 | 196 | 186 | 183 | 964
  White | 1209 | 1200 | 1212 | 1223 | 1223 | 6067
  More than one race | 66 | 64 | 55 | 53 | 66 | 304
  Unknown or Not Reported | 60 | 52 | 51 | 49 | 47 | 259
Education [Count of Participants; unit: Participants]
  High school diploma or less | 417 | 401 | 426 | 437 | 436 | 2117
  Some college | 409 | 361 | 337 | 367 | 340 | 1814
  College graduate or associate degree | 596 | 650 | 639 | 627 | 614 | 3126
  Graduate degree | 171 | 175 | 186 | 159 | 197 | 888

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Purchasing Beverages With Calories
Description: Participants will select a beverage to purchase from the online vending machine. Outcome is binary: purchased a beverage with calories or not.
Time Frame: The survey will take up to 20 minutes.
Population: Participants were excluded from this outcome if a) they requested their data be excluded after being debriefed about the purpose of the study, b) they finished the survey too quickly (i.e., faster than 191.2 seconds which was 1/3 of the median completion time in a soft launch of the survey), or they were missing on this outcome (n=2).
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Green Labels | Traffic Light Labels | Physical Activity Calorie Equivalent Labels | "High in" Nutrient Warning Labels
Number analyzed (Participants) | 1592 | 1587 | 1588 | 1589 | 1587
Participants | 1005 | 765 | 763 | 748 | 847

2. Primary Outcome: Calories Purchased From Beverages, if Beverage With Calories Chosen
Description: Participants will select a beverage to purchase from the online vending machine. Outcome is calories in beverage chosen to purchase - only for those participants who chose a beverage with calories.
Time Frame: The survey will take up to 20 minutes.
Population: Participants were excluded from this outcome if a) they requested their data be excluded after being debriefed about the purpose of the study, b) they finished the survey too quickly (i.e., faster than 191.2 seconds which was 1/3 of the median completion time in a soft launch of the survey), c) they were missing on this outcome (n=2), or d) they did not choose a beverage with calories.
Measure: Mean (Standard Deviation); unit: Beverage calories
Arm/Group | Control | Green Labels | Traffic Light Labels | Physical Activity Calorie Equivalent Labels | "High in" Nutrient Warning Labels
Number analyzed (Participants) | 1005 | 765 | 763 | 748 | 847
Beverage calories | 199 (84) | 190 (90) | 196 (87) | 184 (92) | 183 (93)

3. Primary Outcome: Calories Purchased From Snacks
Description: Participants will select a snack to purchase from the online vending machine. Outcome is calories in snacks chosen to purchase.
Time Frame: The survey will take up to 20 minutes.
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Snack calories
Arm/Group | Control | Green Labels | Traffic Light Labels | Physical Activity Calorie Equivalent Labels | "High in" Nutrient Warning Labels
Number analyzed (Participants) | 1593 | 1587 | 1588 | 1590 | 1587
Snack calories | 183 (69) | 170 (62) | 169 (63) | 164 (68) | 169 (67)

4. Secondary Outcome: Likelihood of Selecting a Healthy Beverage
Description: Participants will select a beverage to purchase in the virtual store. Outcome is percentage of people selecting a healthy beverage (green labeled in the traffic light condition)
Time Frame: The survey will take up to 20 minutes.
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Green Labels | Traffic Light Labels | Physical Activity Calorie Equivalent Labels | "High in" Nutrient Warning Labels
Number analyzed (Participants) | 1592 | 1587 | 1588 | 1589 | 1587
Participants | 311 | 526 | 601 | 473 | 412

5. Secondary Outcome: Likelihood of Selecting a Moderately Healthy Beverage
Description: Participants will select a beverage to purchase in the virtual store. Outcome is percentage of people selecting a moderately healthy beverage (yellow labeled in the traffic light condition)
Time Frame: The survey will take up to 20 minutes.
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Green Labels | Traffic Light Labels | Physical Activity Calorie Equivalent Labels | "High in" Nutrient Warning Labels
Number analyzed (Participants) | 1592 | 1587 | 1588 | 1589 | 1587
Participants | 459 | 471 | 420 | 564 | 549

6. Secondary Outcome: Likelihood of Selecting a Less Healthy Beverage
Description: Participants will select a beverage to purchase in the virtual store. Outcome is percentage of people selecting a less healthy beverage (red labeled in the traffic light condition)
Time Frame: The survey will take up to 20 minutes.
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Green Labels | Traffic Light Labels | Physical Activity Calorie Equivalent Labels | "High in" Nutrient Warning Labels
Number analyzed (Participants) | 1592 | 1587 | 1588 | 1589 | 1587
Participants | 822 | 590 | 567 | 552 | 626

7. Secondary Outcome: Likelihood of Selecting a Healthy Snack
Description: Participants will select a snack to purchase in the virtual store. Outcome is percentage of people selecting a healthy snack (green labeled in the traffic light condition)
Time Frame: The survey will take up to 20 minutes.
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Green Labels | Traffic Light Labels | Physical Activity Calorie Equivalent Labels | "High in" Nutrient Warning Labels
Number analyzed (Participants) | 1593 | 1587 | 1588 | 1590 | 1587
Participants | 268 | 480 | 494 | 384 | 427

8. Secondary Outcome: Likelihood of Selecting a Moderately Healthy Snack
Description: Participants will select a snack to purchase in the virtual store. Outcome is percentage of people selecting a moderately healthy snack (yellow labeled in the traffic light condition)
Time Frame: The survey will take up to 20 minutes.
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Green Labels | Traffic Light Labels | Physical Activity Calorie Equivalent Labels | "High in" Nutrient Warning Labels
Number analyzed (Participants) | 1593 | 1587 | 1588 | 1590 | 1587
Participants | 677 | 619 | 673 | 733 | 706

9. Secondary Outcome: Likelihood of Selecting a Less Healthy Snack
Description: Participants will select a snack to purchase in the virtual store. Outcome is percentage of people selecting a less healthy snack (red labeled in the traffic light condition)
Time Frame: The survey will take up to 20 minutes.
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Green Labels | Traffic Light Labels | Physical Activity Calorie Equivalent Labels | "High in" Nutrient Warning Labels
Number analyzed (Participants) | 1593 | 1587 | 1588 | 1590 | 1587
Participants | 648 | 488 | 421 | 473 | 454

10. Secondary Outcome: Saturated Fat Purchased From Beverages
Description: Participants will select a beverage to purchase from the online vending machine. Outcome is saturated fat in beverage chosen to purchase.
Time Frame: The survey will take up to 20 minutes.
Measure: Mean (Full Range); unit: grams
Arm/Group | Control | Green Labels | Traffic Light Labels | Physical Activity Calorie Equivalent Labels | "High in" Nutrient Warning Labels
Number analyzed (Participants) | 1592 | 1587 | 1588 | 1589 | 1587
grams | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]

11. Secondary Outcome: Sodium Purchased From Beverages
Description: Participants will select a beverage to purchase from the online vending machine. Outcome is sodium in beverage chosen to purchase.
Time Frame: The survey will take up to 20 minutes.
Measure: Mean (Standard Deviation); unit: milligrams
Arm/Group | Control | Green Labels | Traffic Light Labels | Physical Activity Calorie Equivalent Labels | "High in" Nutrient Warning Labels
Number analyzed (Participants) | 1592 | 1587 | 1588 | 1589 | 1587
milligrams | 94 (82) | 81 (85) | 71 (82) | 88 (88) | 93 (88)

12. Secondary Outcome: Total Sugar Purchased From Beverages
Description: Participants will select a beverage to purchase from the online vending machine. Outcome is total sugar in beverage chosen to purchase.
Time Frame: The survey will take up to 20 minutes.
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Control | Green Labels | Traffic Light Labels | Physical Activity Calorie Equivalent Labels | "High in" Nutrient Warning Labels
Number analyzed (Participants) | 1592 | 1587 | 1588 | 1589 | 1587
grams | 33 (31) | 24 (30) | 24 (30) | 22 (30) | 25 (30)

13. Secondary Outcome: Saturated Fat Purchased From Snacks
Description: Participants will select a snack to purchase from the online vending machine. Outcome is saturated fat in snack chosen to purchase.
Time Frame: The survey will take up to 20 minutes.
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Control | Green Labels | Traffic Light Labels | Physical Activity Calorie Equivalent Labels | "High in" Nutrient Warning Labels
Number analyzed (Participants) | 1593 | 1587 | 1588 | 1590 | 1587
grams | 2.2 (1.9) | 1.8 (1.8) | 1.6 (1.7) | 1.7 (1.8) | 1.6 (1.8)

14. Secondary Outcome: Sodium Purchased From Snacks
Description: Participants will select a snack to purchase from the online vending machine. Outcome is sodium in snack chosen to purchase.
Time Frame: The survey will take up to 20 minutes.
Measure: Mean (Standard Deviation); unit: milligrams
Arm/Group | Control | Green Labels | Traffic Light Labels | Physical Activity Calorie Equivalent Labels | "High in" Nutrient Warning Labels
Number analyzed (Participants) | 1593 | 1587 | 1588 | 1590 | 1587
milligrams | 150 (74) | 153 (67) | 153 (68) | 142 (73) | 144 (74)

15. Secondary Outcome: Total Sugar Purchased From Snacks
Description: Participants will select a snack to purchase from the online vending machine. Outcome is total sugar in snack chosen to purchase.
Time Frame: The survey will take up to 20 minutes.
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Control | Green Labels | Traffic Light Labels | Physical Activity Calorie Equivalent Labels | "High in" Nutrient Warning Labels
Number analyzed (Participants) | 1593 | 1587 | 1588 | 1590 | 1587
grams | 12 (14) | 9 (13) | 8 (13) | 9 (13) | 9 (14)

16. Secondary Outcome: Perceived Healthiness of a Healthy Beverage
Description: This variable will be measured on a 5-point Likert scale ranging from "very unhealthy" to "very healthy".
Time Frame: The survey will take up to 20 minutes.
Measure: Mean (Standard Deviation); unit: units on a 1-5 scale
Arm/Group | Control | Green Labels | Traffic Light Labels | Physical Activity Calorie Equivalent Labels | "High in" Nutrient Warning Labels
Number analyzed (Participants) | 1592 | 1587 | 1588 | 1590 | 1587
units on a 1-5 scale | 3.8 (0.9) | 4.0 (0.9) | 4.0 (1.0) | 4.0 (1.0) | 4.0 (1.0)

17. Secondary Outcome: Perceived Healthiness of a Moderately Healthy Beverage
Description: This variable will be measured on a 5-point Likert scale ranging from "very unhealthy" to "very healthy".
Time Frame: The survey will take up to 20 minutes.
Measure: Mean (Standard Deviation); unit: units on a 1-5 scale
Arm/Group | Control | Green Labels | Traffic Light Labels | Physical Activity Calorie Equivalent Labels | "High in" Nutrient Warning Labels
Number analyzed (Participants) | 1593 | 1587 | 1588 | 1590 | 1587
units on a 1-5 scale | 3.7 (1.0) | 3.5 (1.0) | 3.3 (1.0) | 3.6 (1.0) | 3.7 (1.0)

18. Secondary Outcome: Perceived Healthiness of a Less Healthy Beverage
Description: This variable will be measured on a 5-point Likert scale ranging from "very unhealthy" to "very healthy".
Time Frame: The survey will take up to 20 minutes.
Measure: Mean (Standard Deviation); unit: units on a 1-5 scale
Arm/Group | Control | Green Labels | Traffic Light Labels | Physical Activity Calorie Equivalent Labels | "High in" Nutrient Warning Labels
Number analyzed (Participants) | 1593 | 1587 | 1588 | 1590 | 1587
units on a 1-5 scale | 3.4 (1.1) | 3.2 (1.1) | 2.7 (1.2) | 3.0 (1.1) | 2.8 (1.2)

19. Secondary Outcome: Perceived Healthiness of a Healthy Snack
Description: This variable will be measured on a 5-point Likert scale ranging from "very unhealthy" to "very healthy".
Time Frame: The survey will take up to 20 minutes.
Measure: Mean (Standard Deviation); unit: units on a 1-5 scale
Arm/Group | Control | Green Labels | Traffic Light Labels | Physical Activity Calorie Equivalent Labels | "High in" Nutrient Warning Labels
Number analyzed (Participants) | 1593 | 1587 | 1588 | 1590 | 1587
units on a 1-5 scale | 3.3 (1.0) | 3.4 (1.0) | 3.6 (1.1) | 2.9 (1.0) | 3.1 (1.0)

20. Secondary Outcome: Perceived Healthiness of a Moderately Healthy Snack
Description: This variable will be measured on a 5-point Likert scale ranging from "very unhealthy" to "very healthy".
Time Frame: The survey will take up to 20 minutes.
Measure: Mean (Standard Deviation); unit: units on a 1-5 scale
Arm/Group | Control | Green Labels | Traffic Light Labels | Physical Activity Calorie Equivalent Labels | "High in" Nutrient Warning Labels
Number analyzed (Participants) | 1593 | 1587 | 1588 | 1590 | 1587
units on a 1-5 scale | 2.7 (1.0) | 2.7 (1.0) | 2.7 (1.0) | 2.6 (1.0) | 2.4 (1.0)

21. Secondary Outcome: Perceived Healthiness of a Less Healthy Snack
Description: This variable will be measured on a 5-point Likert scale ranging from "very unhealthy" to "very healthy".
Time Frame: The survey will take up to 20 minutes.
Measure: Mean (Standard Deviation); unit: units on a 1-5 scale
Arm/Group | Control | Green Labels | Traffic Light Labels | Physical Activity Calorie Equivalent Labels | "High in" Nutrient Warning Labels
Number analyzed (Participants) | 1593 | 1587 | 1588 | 1588 | 1587
units on a 1-5 scale | 2.3 (1.0) | 2.3 (1.0) | 2.0 (1.0) | 2.2 (1.0) | 2.0 (1.0)

22. Secondary Outcome: Noticing Trial Labels
Description: Participants will respond "yes," "no," or "not sure" to the item: "When you were selecting a beverage and a snack, did you notice any other nutrition labels on or next to the products?"
Time Frame: The survey will take up to 20 minutes.
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Green Labels | Traffic Light Labels | Physical Activity Calorie Equivalent Labels | "High in" Nutrient Warning Labels
Number analyzed (Participants) | 1591 | 1585 | 1585 | 1590 | 1583
Participants
  No | 859 | 675 | 635 | 623 | 459
  Yes | 538 | 692 | 711 | 772 | 960
  Not sure | 194 | 218 | 239 | 195 | 164

23. Secondary Outcome: Degree of Perceived Label Influence on Beverage Selection
Description: Participants will respond on a 5-point scale ranging from "Not at all" to "A great deal" to the item: "How much did you use this label to help you decide what beverage to buy?"
Time Frame: The survey will take up to 20 minutes.
Measure: Mean (Standard Deviation); unit: units on a 1-5 scale
Arm/Group | Control | Green Labels | Traffic Light Labels | Physical Activity Calorie Equivalent Labels | "High in" Nutrient Warning Labels
Number analyzed (Participants) | 1593 | 1587 | 1588 | 1590 | 1587
units on a 1-5 scale | 2.6 (1.3) | 2.4 (1.3) | 2.6 (1.3) | 2.8 (1.4) | 3.0 (1.4)

24. Secondary Outcome: Degree of Perceived Label Influence on Snack Selection
Description: Participants will respond on a 5-point scale ranging from "Not at all" to "A great deal" to the item: "How much did you use this label to help you decide what snack to buy?"
Time Frame: The survey will take up to 20 minutes.
Measure: Mean (Standard Deviation); unit: units on a 1-5 scale
Arm/Group | Control | Green Labels | Traffic Light Labels | Physical Activity Calorie Equivalent Labels | "High in" Nutrient Warning Labels
Number analyzed (Participants) | 1593 | 1587 | 1588 | 1590 | 1587
units on a 1-5 scale | 2.4 (1.3) | 2.4 (1.3) | 2.6 (1.3) | 2.8 (1.4) | 3.0 (1.4)

25. Secondary Outcome: Trust in Labels
Description: Item: "How much do you trust or distrust the information on this label?". Responses will be measured on a 5-point Likert scale from "completely distrust" to "completely trust".
Time Frame: The survey will take up to 20 minutes.
Measure: Mean (Standard Deviation); unit: units on a 1-5 scale
Arm/Group | Control | Green Labels | Traffic Light Labels | Physical Activity Calorie Equivalent Labels | "High in" Nutrient Warning Labels
Number analyzed (Participants) | 1593 | 1587 | 1588 | 1590 | 1587
units on a 1-5 scale | 3.8 (1.0) | 3.5 (0.9) | 3.6 (1.0) | 3.7 (0.9) | 3.8 (0.9)

26. Secondary Outcome: Reactance to Labels
Description: We will examine the average reactance to the label (said the label is trying to manipulate me, or annoys me). Each reactance item will be scored on a 5-pt likert scale from "not at all" to "a great deal".
Time Frame: The survey will take up to 20 minutes.
Measure: Mean (Standard Deviation); unit: units on a 1-5 scale
Arm/Group | Control | Green Labels | Traffic Light Labels | Physical Activity Calorie Equivalent Labels | "High in" Nutrient Warning Labels
Number analyzed (Participants) | 1593 | 1587 | 1588 | 1590 | 1587
units on a 1-5 scale | 1.9 (1.0) | 2.0 (1.1) | 2.2 (1.1) | 2.0 (1.1) | 2.1 (1.1)

27. Secondary Outcome: Attention to Labels
Description: Item: "How much does this label grab your attention?". Responses will be measured on a 5-point Likert scale from "not at all" to "a great deal".
Time Frame: The survey will take up to 20 minutes.
Measure: Mean (Standard Deviation); unit: units on a 1-5 scale
Arm/Group | Control | Green Labels | Traffic Light Labels | Physical Activity Calorie Equivalent Labels | "High in" Nutrient Warning Labels
Number analyzed (Participants) | 1593 | 1587 | 1588 | 1590 | 1586
units on a 1-5 scale | 3.3 (1.2) | 3.2 (1.2) | 3.4 (1.2) | 3.5 (1.2) | 3.5 (1.2)

28. Secondary Outcome: Learned From Labels
Description: Item: "To what extent did you learn something new from this label?". Responses will be measured on a 5-point Likert scale from "not at all" to "a great deal".
Time Frame: The survey will take up to 20 minutes.
Measure: Mean (Standard Deviation); unit: units on a 1-5 scale
Arm/Group | Control | Green Labels | Traffic Light Labels | Physical Activity Calorie Equivalent Labels | "High in" Nutrient Warning Labels
Number analyzed (Participants) | 1593 | 1587 | 1588 | 1590 | 1587
units on a 1-5 scale | 2.7 (1.2) | 2.8 (1.3) | 3.1 (1.2) | 3.5 (1.2) | 3.2 (1.2)

29. Secondary Outcome: Thinking About Health Effects
Description: Item: "How much does this label make you think about the health effects of food and beverages?". Responses will be measured on a 5-point Likert scale from "not at all" to "a great deal"
Time Frame: The survey will take up to 20 minutes.
Measure: Mean (Standard Deviation); unit: units on a 1-5 scale
Arm/Group | Control | Green Labels | Traffic Light Labels | Physical Activity Calorie Equivalent Labels | "High in" Nutrient Warning Labels
Number analyzed (Participants) | 1593 | 1587 | 1588 | 1590 | 1587
units on a 1-5 scale | 3.2 (1.2) | 3.0 (1.3) | 3.3 (1.2) | 3.4 (1.3) | 3.5 (1.2)

30. Secondary Outcome: Perceived Discouragement
Description: We will examine if they said the label discourages them from choosing unhealthy products. This item will be scored on a 5-pt likert scale from "not at all" to "a great deal"
Time Frame: The survey will take up to 20 minutes.
Measure: Mean (Standard Deviation); unit: units on a 1-5 scale
Arm/Group | Control | Green Labels | Traffic Light Labels | Physical Activity Calorie Equivalent Labels | "High in" Nutrient Warning Labels
Number analyzed (Participants) | 1593 | 1586 | 1588 | 1589 | 1587
units on a 1-5 scale | 2.7 (1.3) | 2.5 (1.3) | 2.9 (1.3) | 3.1 (1.3) | 3.2 (1.3)

31. Secondary Outcome: Perceived Encouragement
Description: We will examine if they said the label encourages them to choose healthy products. This item will be scored on a 5-pt likert scale from "not at all" to "a great deal"
Time Frame: The survey will take up to 20 minutes.
Measure: Mean (Standard Deviation); unit: units on a 1-5 scale
Arm/Group | Control | Green Labels | Traffic Light Labels | Physical Activity Calorie Equivalent Labels | "High in" Nutrient Warning Labels
Number analyzed (Participants) | 1593 | 1586 | 1588 | 1590 | 1587
units on a 1-5 scale | 3.0 (1.3) | 3.0 (1.3) | 3.2 (1.3) | 3.3 (1.3) | 3.3 (1.3)

32. Secondary Outcome: Negative Emotional Reactions
Description: We will examine the average negative emotional response to the label (said the label made them feel worried, scared, guilty, ashamed, or sad). Each emotion will be scored on a 5-pt likert scale from "not at all" to "a great deal".
Time Frame: The survey will take up to 20 minutes.
Measure: Mean (Standard Deviation); unit: units on a 1-5 scale
Arm/Group | Control | Green Labels | Traffic Light Labels | Physical Activity Calorie Equivalent Labels | "High in" Nutrient Warning Labels
Number analyzed (Participants) | 1592 | 1587 | 1588 | 1590 | 1587
units on a 1-5 scale | 1.7 (0.9) | 1.5 (0.8) | 1.8 (0.9) | 1.9 (1.0) | 2.0 (1.0)

33. Secondary Outcome: Perceived Control in Response to Labels
Description: Participants will respond to the item "Overall does this label make you feel…" with one of 3 responses: "less in control of making healthy eating decisions", "more in control of healthy eating decisions", or "neither less nor more in control of making healthy eating decisions"
Time Frame: The survey will take up to 20 minutes.
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Green Labels | Traffic Light Labels | Physical Activity Calorie Equivalent Labels | "High in" Nutrient Warning Labels
Number analyzed (Participants) | 1593 | 1586 | 1588 | 1589 | 1587
Participants
  Decreased control | 82 | 55 | 60 | 80 | 60
  Neither decrease/increase | 769 | 872 | 757 | 644 | 611
  Increased control | 742 | 659 | 771 | 865 | 916

34. Secondary Outcome: Perceived Personal Stigmatization
Description: Participants will respond to the item "How personally stigmatized does this label make you feel?" on a 5-pt likert scale from "not at all" to "a great deal".
Time Frame: The survey will take up to 20 minutes.
Measure: Mean (Standard Deviation); unit: units on a 1-5 scale
Arm/Group | Control | Green Labels | Traffic Light Labels | Physical Activity Calorie Equivalent Labels | "High in" Nutrient Warning Labels
Number analyzed (Participants) | 1593 | 1587 | 1588 | 1589 | 1587
units on a 1-5 scale | 1.9 (1.2) | 1.8 (1.1) | 2.1 (1.2) | 2.0 (1.2) | 2.1 (1.2)

35. Secondary Outcome: Perceived Obesity Stigma
Description: We will examine the average stigma response to the label (the label stigmatizes people with obesity, the label increases blame toward people for being overweight). Each stigma item will be scored on a 5-pt likert scale from "not at all" to "a great deal".
Time Frame: The survey will take up to 20 minutes.
Measure: Mean (Standard Deviation); unit: units on a 1-5 scale
Arm/Group | Control | Green Labels | Traffic Light Labels | Physical Activity Calorie Equivalent Labels | "High in" Nutrient Warning Labels
Number analyzed (Participants) | 1593 | 1587 | 1588 | 1590 | 1587
units on a 1-5 scale | 2.1 (1.2) | 1.9 (1.1) | 2.3 (1.2) | 2.2 (1.2) | 2.4 (1.2)

36. Secondary Outcome: Disgust Toward People With Obesity
Description: Participants will respond to the item "How disgusted do people with obesity make you feel?" on a 5-pt likert scale from "not at all" to "a great deal".
Time Frame: The survey will take up to 20 minutes.
Measure: Mean (Standard Deviation); unit: units on a 1-5 scale
Arm/Group | Control | Green Labels | Traffic Light Labels | Physical Activity Calorie Equivalent Labels | "High in" Nutrient Warning Labels
Number analyzed (Participants) | 1593 | 1586 | 1588 | 1590 | 1587
units on a 1-5 scale | 2.0 (1.2) | 1.9 (1.2) | 2.0 (1.1) | 1.9 (1.2) | 2.0 (1.2)

ADVERSE EVENTS:
Time Frame: 20 minutes
Arm/Group | Control | Green Labels | Traffic Light Labels | Physical Activity Calorie Equivalent Labels | "High in" Nutrient Warning Labels
All-Cause Mortality (participants affected / at risk) | 0/1627 | 0/1639 | 0/1623 | 0/1633 | 0/1623
Serious Adverse Events (participants affected / at risk) | 0/1627 | 0/1639 | 0/1623 | 0/1633 | 0/1623
Other Adverse Events (participants affected / at risk) | 0/1627 | 0/1639 | 0/1623 | 0/1633 | 0/1623

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-31): https://cdn.clinicaltrials.gov/large-docs/71/NCT05432271/Prot_SAP_000.pdf